CLINICAL TRIAL: NCT05099601
Title: Topical Silymarin Versus Combined Topical Silymarin and Microneedling in Treatment of Melasma: Split Face Study
Brief Title: Silymarin Cream Versus Combined Silymarin Cream and Microneedling in Treatment of Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Abd El-nasser Attay, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSM
Record Dates: First submitted 2021-10-02; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Silymarin; Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Each side of the patients' face will be randomly allocated to either topical silymarin 0.7% and microneedling or topical silymarin 0.7% alone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silymarin alone versus silymarin and microneedling (Experimental): There will be one group of patients. Each side of the patients' face will be randomly allocated to either topical silymarin 0.7% and microneedling or topical silymarin 0.7% alone.
  Interventions: Combination Product: Silymarin; Procedure: Microneedling

INTERVENTIONS:
Combination Product: Silymarin — The patients will use topical silymarin 0.7% cream on the face twice daily(home use).
Procedure: Microneedling — Patients will be subjected to microneedling sessions on one side of the face. Three consecutive sessions, 4 weeks apart (0, 4, 8 weeks), will be performed by dermapen. Sessions will be done by well trained physician.

SUMMARY:
Melasma is an acquired pigmentary disorder, occurring most commonly on the face. It is more prevalent in females and darker skin types. Melasma is mainly a clinical diagnosis consisting of symmetric reticulated hypermelanosis in three predominant facial patterns: centrofacial, malar, and mandibular. Melasma, though benign, can be extremely psychologically distressing and has been shown to have a significant impact on quality of life, social and emotional wellbeing. Multiple factors are implicated in the pathogenesis of melasma; however, the definite underlying mechanisms are not yet completely established. Ultraviolet exposure is one of the leading etiological factors, besides genetic and hormonal factors.

DETAILED DESCRIPTION:
Many studies examined multiple treatment options for melasma, but none of them is completely satisfactory with recurrence in most cases.

Silymarin (SM) is a standardized extract from Silybum marianum seeds, is traditionally used as a hepatoprotective agent for its potent regenerative properties. Lately, SM is utilized in dermatological and cosmetic preparations for its antioxidant effect, anti-inflammatory and immunomodulatory properties.

Silibinin, the main component of silymarin, has been found to have antioxidant properties. It decreases the hazardous effects of solar ultraviolet radiation and significantly prevents melanin production in a dose-dependent manner without effect on cell viability.

Skin microneedling, or percutaneous collagen induction by needles, is a minimally invasive procedure that uses short fine needles to puncture the skin and stimulates fibroblast proliferation, release of growth factors and collagen production.

Long-term improvement of melasma after microneedling was reported , however, the exact mechanism that promotes skin lightening is not known.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years old.
* Pattern of melasma: Bilateral symmetrical facial melasma of any pattern.
* Fitzpatrick skin phototypes: Types III, IV and V

Exclusion Criteria:

* Pregnancy and lactation.
* Patients taking oral contraceptive pills, hormonal replacement therapy or treatment for chronic illness at the time of the study or during the past 6 months.
* Coexistance of diseases associated with hyperpigmentation such as Addison disease.
* Scarring and keloid tendency, active skin infections as active HSV.
* Previous history of post inflammatory hyperpigmentation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
compare between the efficacy of topical silymarin alone and its combination with microneedling in treatment of melasma. | 3 months
  Scoring of the patients according to modified Melasma Area and Severity Index (mMASI) score before and after treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balkrishnan R, McMichael AJ, Camacho FT, Saltzberg F, Housman TS, Grummer S, Feldman SR, Chren MM. Development and validation of a health-related quality of life instrument for women with melasma. Br J Dermatol. 2003 Sep;149(3):572-7. doi: 10.1046/j.1365-2133.2003.05419.x. PMID 14510991
- [Background] Choo SJ, Ryoo IJ, Kim YH, Xu GH, Kim WG, Kim KH, Moon SJ, Son ED, Bae K, Yoo ID. Silymarin inhibits melanin synthesis in melanocyte cells. J Pharm Pharmacol. 2009 May;61(5):663-7. doi: 10.1211/jpp/61.05.0016. PMID 19406006
- [Background] Cohen BE, Elbuluk N. Microneedling in skin of color: A review of uses and efficacy. J Am Acad Dermatol. 2016 Feb;74(2):348-55. doi: 10.1016/j.jaad.2015.09.024. PMID 26549251
- [Background] Handel AC, Miot LD, Miot HA. Melasma: a clinical and epidemiological review. An Bras Dermatol. 2014 Sep-Oct;89(5):771-82. doi: 10.1590/abd1806-4841.20143063. PMID 25184917
- [Background] Hou A, Cohen B, Haimovic A, Elbuluk N. Microneedling: A Comprehensive Review. Dermatol Surg. 2017 Mar;43(3):321-339. doi: 10.1097/DSS.0000000000000924. PMID 27755171
- [Background] Kimbrough-Green CK, Griffiths CE, Finkel LJ, Hamilton TA, Bulengo-Ransby SM, Ellis CN, Voorhees JJ. Topical retinoic acid (tretinoin) for melasma in black patients. A vehicle-controlled clinical trial. Arch Dermatol. 1994 Jun;130(6):727-33. PMID 8002642
- [Background] Kren V, Walterova D. Silybin and silymarin--new effects and applications. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2005 Jun;149(1):29-41. doi: 10.5507/bp.2005.002. PMID 16170386
- [Background] Nofal A, Ibrahim AM, Nofal E, Gamal N, Osman S. Topical silymarin versus hydroquinone in the treatment of melasma: A comparative study. J Cosmet Dermatol. 2019 Feb;18(1):263-270. doi: 10.1111/jocd.12769. Epub 2018 Aug 26. PMID 30146802
- [Background] Pandya AG, Hynan LS, Bhore R, Riley FC, Guevara IL, Grimes P, Nordlund JJ, Rendon M, Taylor S, Gottschalk RW, Agim NG, Ortonne JP. Reliability assessment and validation of the Melasma Area and Severity Index (MASI) and a new modified MASI scoring method. J Am Acad Dermatol. 2011 Jan;64(1):78-83, 83.e1-2. doi: 10.1016/j.jaad.2009.10.051. Epub 2010 Apr 15. PMID 20398960
- [Background] Rigopoulos D, Gregoriou S, Katsambas A. Hyperpigmentation and melasma. J Cosmet Dermatol. 2007 Sep;6(3):195-202. doi: 10.1111/j.1473-2165.2007.00321.x. PMID 17760699
- [Background] Tamega Ade A, Miot LD, Bonfietti C, Gige TC, Marques ME, Miot HA. Clinical patterns and epidemiological characteristics of facial melasma in Brazilian women. J Eur Acad Dermatol Venereol. 2013 Feb;27(2):151-6. doi: 10.1111/j.1468-3083.2011.04430.x. Epub 2012 Jan 3. PMID 22212073
- [Background] Tran JM, Chan AW (2012) Quick diagnosis: melasma. University of Toronto Med J 89: 143-145.
- [Background] Vaid M, Katiyar SK. Molecular mechanisms of inhibition of photocarcinogenesis by silymarin, a phytochemical from milk thistle (Silybum marianum L. Gaertn.) (Review). Int J Oncol. 2010 May;36(5):1053-60. doi: 10.3892/ijo_00000586. PMID 20372777
- [Background] Wu DC, Fitzpatrick RE, Goldman MP. Confetti-like Sparing: A Diagnostic Clinical Feature of Melasma. J Clin Aesthet Dermatol. 2016 Feb;9(2):48-57. PMID 27047632